CLINICAL TRIAL: NCT03846921
Title: Alpha-defensin as a Diagnostic Means to Distinguish Between Acute Bacterial and Viral Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0003-19
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-02

CONDITIONS: Bacterial Infections; Viral Infection
MeSH Terms: conditions — Bacterial Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Viral infection: Patients with proven viral infections will have laboratory blood test taken
  Interventions: Diagnostic Test: Laboratory blood test
- Bacterial Infection: Patients with proven bacterial infections will have laboratory blood test taken
  Interventions: Diagnostic Test: Laboratory blood test

INTERVENTIONS:
Diagnostic Test: Laboratory blood test — Laboratory blood test will be analyzed to determine whether there is a rise in alpha-defensin

SUMMARY:
This study aims to investigate the use of alpha-defensin as a diagnostic means to distinguish between acute bacterial and viral infections.

ELIGIBILITY:
Inclusion Criteria:

* Children with either bacterial or viral infections

Exclusion Criteria:

* All others

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with fever attending pediatric emergency department or who have been hospitalized
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Rise in alpha-defensin | One year
  Laboratory blood tests will be analyzed to determine whether there is a rise in alpha-defensin levels in bacterial infections as compared to viral infections.

CONTACTS AND LOCATIONS:
Overall Officials: Eias Kassem, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No